CLINICAL TRIAL: NCT03565432
Title: Sick Leave, Work Disability and Quality of Life in Korean Patients With Inflammatory Bowel Diseases : A Prospective Survey Study
Brief Title: Sick Leave, Work Disability and Quality of Life in Korean Patients With Inflammatory Bowel Diseases
Status: Completed | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Professor, Kyunghee University Medical Center
Other Study IDs: IBDWORK2018
Record Dates: First submitted 2018-04-25; First posted 2018-06-21 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: work disability; quality of life; psychosocial distress
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD in KHUH: Registered patients with Inflammatory bowel disease at Kyung Hee University Hospital

SUMMARY:
Inflammatory bowel diseases (IBD) is a chronic inflammatory condition of the gastrointestinal tract that significantly affects quality of life of patients.

Several studies have reported that the loss of work productivity is significantly higher than that of the general population due to disease-related symptoms and various factors in patients with inflammatory bowel disease in Western countries, but there is few data in Korea.

Therefore, this study is to assess the effect of disease on sick leave, work disability and health related quality of life in Korean patients with inflammatory bowel disease by using validated questionnaires.

DETAILED DESCRIPTION:
First, the investigators will estimate the prevalence of work disability in patients with inflammatory bowel disease using the Work Productivity and Activity Index (WPAI), that have been validated in patients with inflammatory bowel disease.

Secondary, the predictor of work productivity impairment in patients with inflammatory bowel disease and distribution of type and severity of work disability will be identified.

Third, the investigators will explore the correlation between the quality of life and psychosocial aspects (anxiety disorder, depression) of patients with inflammatory bowel disease.

One year later, the same questionnaire will be surveyed repeatedly in the same participants under usual care to investigate the changes in patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with inflammatory bowel disease (Crohn's disease and ulcerative colitis) at Kyung Hee University Hospital

Exclusion Criteria:

1. Patients who do not agree to fill out the questionnaire.
2. Patients who can not fill out the questionnaire themselves.
3. Patients who can not understand the questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with inflammatory bowel disease (Crohn disease and ulcerative colitis) at Kyung Hee University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Mean Total Percentage of Work Impairment by Work Productivity and Activity Impairment Questionnaire (WPAI) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The WPAI assess the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI includes 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answer questions related to employment status and activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity
Mean Work Time Missed by WPAI in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The WPAI assess the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI includes 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answer questions related to employment status and activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity.
Mean Impairment while Working by WPAI in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The WPAI assess the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI includes 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answer questions related to employment status and activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity
Mean Total Activity Impairment by WPAI in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The WPAI assess the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI includes 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answer questions related to employment status and activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity.

SECONDARY OUTCOMES:
Mean Score of Crohn's and ulcerative colitis Questionnaire-8 (CUCQ-8) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The investigator will estimate the disease specific quality of life in patients with ulcerative colitis or crohn disease, using validated questionnaires - Crohn's and ulcerative colitis Questionnaire-8 (CUCQ-8).
  CUCQ-8 : total score is evaluated from 0 (greatest QoL) to 24 (poorest QoL) with each items scoring range from 0 to 3
Mean Score of and inflammatory Bowel Disease Disability Index (IBD-DI) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The investigator will estimate the disability in patients with ulcerative colitis or crohn disease, using validated questionnaire inflammatory Bowel Disease Disability Index (IBD-DI) IBD-DI : Each item is rated at 1-5 and interpretated for disability at -80 (maximum degree of disability) to 22 (no disability).
Mean Score of Hospital Anxiety and Depression Scale (HADS) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The investigators will evaluate the prevalence and severity of psychosocial distress (anxiety and depression disorder) using variable validated questionnaires that Hospital Anxiety and Depression Scale HADS : Scores are interpreted as 0-7: normal, 8-10: borderline, 11-21: significant and the higher score means the more significant psychosocial distress.
Mean Score of Patient Health Questionnaire-9 (PHQ-9) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The investigators will evaluate the prevalence and severity of psychosocial distress (anxiety and depression disorder) using variable validated questionnaires that Patient Health Questionnaire-9 (PHQ-9).
  PHQ-9 : 0-4: minimal, 5-9: mild,10-14: moderate,15-19: moderately severe, 20-27: Severe, and 10 points or more are interpreted as major depression.
Mean Score of Anxious thoughts and tendencies (AT&T) in CD or UC Participants | From initial diagnosis until date of data collection (approximately 1 years)
  The investigators will evaluate the prevalence and severity of anxiety disorder using variable validated questionnaires that Anxious thoughts and tendencies (AT&T).
  AT&T:Based on the degree of anxiety, the total score is calculated from 4 points to 60 points.The higher score means the more significant anxiety disorder.

OTHER OUTCOMES:
Correlation between work disability, psychosocial distress and quality of life | From initial diagnosis until date of data collection (approximately 1 years)
  Pearson coefficient analysis will be used to analyze the correlations between the results of each questionnaire (psychosocial distress, Quality of life and work disability) And two or three of outcomes with higher correlation efficient will be re-analyzed after adjustment of each variables.
Predictors that cause a decrease in work productivity of patients with inflammatory bowel disease | From initial diagnosis until date of data collection (approximately 1 years)
  Predictors that may cause a decrease in work productivity of patients with inflammatory bowel disease will identified using linear regression analysis of multiple baseline variables and the score from Work productivity and Activity Index (WPAI) questionnaire.
Mean Change From Baseline in Work Productivity and Activity Impairment (WPAI) under usual care at Year1 | From initial diagnosis until date of data collection (approximately 1 years)
  The WPAI assess the impact of IBD on work productivity and daily activities during the previous 7 days. The WPAI includes 6 questions: 1 (if currently employed); 2 (hours missed due to disease); 3 (hours missed other reasons); 4 (hours actually worked); 5 (degree disease affected productivity while working); 6 (degree disease affected regular activities). WPAI generates four component scores: percentage of work time missed (absenteeism); percentage of impairment while working (presentisms); percentage of overall work impairment (absenteeism and presentisms combined); and percentage of activity impairment. Unemployed participants only answer questions related to employment status and activity impairment. Scores for WPAI range from 0% to 100%, where 0 % indicates no impairment and 100% is total loss of work productivity/activity
Mean Change From Baseline in Crohn's and ulcerative colitis Questionnaire-8 (CUCQ-8) under usual care at Year1. | From initial diagnosis until date of data collection (approximately 1 years)
  CUCQ-8 : total score is evaluated from 0 (greatest QoL) to 24 (poorest QoL) with each items scoring range from 0 to 3.
Mean Change From Baseline in inflammatory Bowel Disease Disability Index (IBD-DI) under usual care at Year1. | From initial diagnosis until date of data collection (approximately 1 years)
  IBD-DI : Each item is rated at 1-5 and interpretated for disability at -80 (maximum degree of disability) to 22 (no disability).
Mean Change From Baseline in Hospital Anxiety and Depression Scale (HADS) under usual care at Year1. | From initial diagnosis until date of data collection (approximately 1 years)
  HADS : Scores are interpreted as 0-7: normal, 8-10: borderline, 11-21: significant and the higher score means the more significant psychosocial distress.
Mean Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) under usual care at Year1 | From initial diagnosis until date of data collection (approximately 1 years)
  PHQ-9 : 0-4: minimal, 5-9: mild,10-14: moderate,15-19: moderately severe, 20-27: Severe, and 10 points or more are interpreted as major depression.
Mean Change From Baseline in Anxious thoughts and tendencies (AT&T) under usual care at Year1 | From initial diagnosis until date of data collection (approximately 1 years)
  AT&T:Based on the degree of anxiety, the total score is calculated from 4 points to 60 points.The higher score means the more significant anxiety disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Kyun Lee, Professor, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
After publishing the results, any data sharing request from other researchers will be positively considered.
  But extent of sharing is not decided yet

REFERENCES:
- [Background] De Boer AG, Bennebroek Evertsz' F, Stokkers PC, Bockting CL, Sanderman R, Hommes DW, Sprangers MA, Frings-Dresen MH. Employment status, difficulties at work and quality of life in inflammatory bowel disease patients. Eur J Gastroenterol Hepatol. 2016 Oct;28(10):1130-6. doi: 10.1097/MEG.0000000000000685. PMID 27340897
- [Background] Vester-Andersen MK, Prosberg MV, Vind I, Andersson M, Jess T, Bendtsen F. Low Risk of Unemployment, Sick Leave, and Work Disability Among Patients with Inflammatory Bowel Disease: A 7-year Follow-up Study of a Danish Inception Cohort. Inflamm Bowel Dis. 2015 Oct;21(10):2296-303. doi: 10.1097/MIB.0000000000000493. PMID 26164663
- [Background] Siebert U, Wurm J, Gothe RM, Arvandi M, Vavricka SR, von Kanel R, Begre S, Sulz MC, Meyenberger C, Sagmeister M; Swiss IBD Cohort Study Group. Predictors of temporary and permanent work disability in patients with inflammatory bowel disease: results of the swiss inflammatory bowel disease cohort study. Inflamm Bowel Dis. 2013 Mar-Apr;19(4):847-55. doi: 10.1097/MIB.0b013e31827f278e. PMID 23446333